CLINICAL TRIAL: NCT01376141
Title: Drug Use Investigation for IMIGRAN Tablet
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 112324
Record Dates: First submitted 2011-03-03; First posted 2011-06-20 (Estimated); Last update posted 2017-05-22 (Actual); Status verified 2017-05

CONDITIONS: Migraine Disorders
MeSH Terms: conditions — Migraine Disorders | interventions — Sumatriptan

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects prescribed IMIGRAN: Subjects with migraine disorders prescribed IMIGRAN during study period
  Interventions: Drug: Sumatriptan

INTERVENTIONS:
Drug: Sumatriptan

SUMMARY:
The study is designed to detect adverse drug reactions (particularly clinically significant adverse drug reactions) occurring in clinical settings, to examine factors likely to affect the safety and efficacy of sumatriptan tablet, and to discuss the need of special investigation and postmarketing clinical study.

A special focus was placed on the investigation of occurrence of "ischaemic heart disease-like events including arrhythmia, angina pectoris, and myocardial infarction" in the present study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with migraine disorders

Exclusion Criteria:

* Subjects with hypersensitivity to sumatriptan
* Subjects with history, symptoms, or signs of myocardial infarction, ischemic cardiac disease, or variant angina
* Subjects with history of peripheral vascular disorder
* Subjects with history of cerebrovascular disorder or transient ischemic attacks
* Subjects with uncontrolled high-blood pressure
* Subjects with severe hepatic function disorder
* Subjects taking ergotamine, ergotamine derivative containing product, or 5-HT1B/1D agonist
* Subjects taking monoamine oxidaze inhibitor or use within 2 weeks of discontinuation

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Male and female Japanese subjects with migraine disorders who were considered appropriate to prescribe sumatriptan tablet according to the prescribing information were eligible for this surveillance study.
Sampling Method: Probability Sample
Enrollment: 3571 (Actual)
Dates: Start 2001-09; Primary Completion 2005-02 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
The number of incidence of adverse events in subjects with migraine disorders | 2 months
  Adverse event (AE), diagnosis or symptom, date of onset, outcome, date of outcome, seriousness, reason for judgement of "serious", intensity, relationship to IMIGRAN, other factors suspected to have relationship to AE

SECONDARY OUTCOMES:
Occurrence of arrhythmia | 2 months
  Occurrence of arrhythmia is investigated throughout study period.
Occurrence of angina pectoris | 2 months
  Occurrence of angina pectoris is investigated throughout study period.
Occurrence of myocardial infarction | 2 months
  Occurrence of myocardial infarction is investigated throughout study period.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline